CLINICAL TRIAL: NCT04769895
Title: Evaluation of the Efficacy of MaaT013 As Salvage Therapy in Acute GVHD Patients with Gastrointestinal Involvement, Refractory to Ruxolitinib; a Multi-center Open-label Phase III Trial.
Brief Title: MaaT013 As Salvage Therapy in Ruxolitinib Refractory GI-aGVHD Patients
Acronym: ARES
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: MaaT Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MPOH06
Record Dates: First submitted 2021-02-22; First posted 2021-02-25 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Acute Graft Versus Host Disease in Intestine; Steroid Refractory GVHD
Keywords: Microbiotherapy; Fecal microbiota transfer; Gastro intestinal acute GVHD; ruxolinib refractory

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MaaT013 (Experimental): Route of administration: rectal (enema)
  Study drug dose: 4 enemas in total:
  Week 1:
  * D0-D1: vancomycin pre-treatment (250mg per os, 4 times a day for 2 days)
  * D2: 1 dose
  * Between D3 to D5: 1 dose Week 2: 1 dose (7 +/- 2 days after the last dose) Week 3: 1 dose (7 +/- 2 days after the last dose) A supplementary dose can be prescribed in case of GvHD relapse or massive antibiotic use during the study.
  Interventions: Drug: MaaT013

INTERVENTIONS:
Drug: MaaT013 — MaaT013 is made of allogeneic, full-ecosystem pooled biotherapeutic intestinal microbiota

SUMMARY:
MaaT013 showed interesting results in steroids and ruxolitinib-resistant aGVHD patients with gut involvement (55% ORR at D28) and 47% and 39% OS at 6 and 12 months respectively (Malard 2020), therefore warrant being tested as salvage therapy in steroid and JAK inhibitors-resistant GI-aGvHD patients. Given the absence of an approved 3rd line strategy or 2nd line strategy in ruxolitinib intolerant patients and the extremely poor prognosis of these patients, who are mostly left with no viable therapeutic option, a single-arm open-label design was proposed.

DETAILED DESCRIPTION:
Standard first-line therapy for the treatment of acute GVHD involves corticosteroids, usually methyl-prednisolone at a dose of 2 mg/kg per day (Martin PJ R. J., 2012; Van Lint MT, 1998). Despite initial responses (around 60%), fewer than half of patients have durable complete responses, and those patients who do not respond or progress after an initial response have high mortality (Weisdorf D, 1990; Alousi AM, 2009; Bolanos-Meade J, 2014). Moreover, prolonged high-dose corticosteroids (CS) exposure is associated with deleterious complications and long-term morbidity (Mohty M, 2010).

For these reasons, there is great interest in identifying effective therapies for corticosteroid-resistant aGvHD and improve outcomes.

Recently, ruxolitinib (Jakafi®), which has an Orphan Drug status in the USA, was granted an approval on 24 May 2019 from the FDA based on study INCB 18424-271 (NCT02953678). This open-label, single-arm study enrolled 72 grade 2-4 SR-aGvHD patients who were treated with 5 mg (possibly increased to 10mg) ruxolitinib b.d. Of the 72 patients, 49 were included in the efficacy evaluation that led the FDA to grant market authorization. Of these 49 patients, Overall Response Rate (ORR - Complete + Very Good Partial + Partial Responses) after 28 days was 100%, 40.7% and 44.4% for patients with Grade 2, Grade 3, and Grade 4 aGVHD respectively. The overall survival (OS) estimate at 6 months was 51.0% for the entire cohort.

The more recent REACH2 phase 3 randomized trial (NCT02913261) investigating ruxolitinib versus best available therapy in patients with corticosteroid-refractory acute GVHD has further established the role of ruxolitinib in the treatment of corticosteroid-refractory acute GvHD. The ORR at day 28 was higher in the ruxolitinib than in the control group (62% versus 39%; odds ratio, 2.64; 95%CI, 1.65-4.22; P<0.001). Similarly, the durable overall response at day 56 was higher in the ruxolitinib than in the control group (40% versus 22%; odds ratio, 2.38; 95% CI, 1.43-3.94; P<0.001) (Zeiser R, 2020) In the REACH1 and REACH2 trials, 45% and 38% of patients, failed to respond to ruxolitinib at day 28, respectively. Moreover, in the REACH2 trial, the overall response at day 56 after initiation of therapy decreased from 62.3% at D28 after initiation of therapy to 39.4% at D56, suggesting a clear unmet medical need for those patients who failed to respond at D28, or worsened afterwards (Zeiser R. 2020). More importantly, results from the REACH1 trial showed only a 22% probability of survival at 2 months in ruxolitinib-non responder patients (Jagasia 2020).

MaaT013 is made of allogeneic, full-ecosystem pooled biotherapeutic intestinal microbiota manufactured by MaaT Pharma in Lyon, France, according to GMP requirements. The intestinal microbiota material in its natural environment is derived from healthy, strictly-vetted and selected donors, following the European consensus recommendations (Cammarota 2016) with the purpose of minimizing the risk associated with fecal material transplants (FMT) for clinical research. Thus, prior to donation, donors undergo a thorough medical evaluation and laboratory screening including SARS-CoV-2 detection, to avoid any known contamination risk. MaaT013 is administered as an enema.

MaaT013 showed interesting results in steroids and ruxolitinib-resistant aGVHD patients with gut involvement (55% ORR at D28) and 47% and 39% OS at 6 and 12 months respectively (Malard 2020), therefore warrant being tested as salvage therapy in steroid and JAK inhibitors-resistant GI-aGvHD patients. Given the absence of an approved 3rd line strategy or 2nd line strategy in ruxolitinib intolerant patients and the extremely poor prognosis of these patients, who are mostly left with no viable therapeutic option, a single-arm open-label design was proposed.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Allo-HSCT with any type of donor, stem cell source, GVHD prophylaxis or conditioning regimen.
* Acute GvHD episode with GI involvement per MAGIC guidelines (= grades II to IV), with or without involvement of other organs
* Patients resistant to steroids AND either resistant to OR with intolerance to ruxolitinib OR with contra-indication to ruxolitinib:

Exclusion Criteria:

* Patients with known hypersensitivity to vancomycin or to any of the excipients listed in the corresponding SmPC
* Patients with active CMV colitis
* Patients who had previously received other lines of systemic aGvHD treatment other than CS and ruxolitinib.
* Grade II-IV hyper-acute GvHD
* Overlap chronic GvHD
* Relapsed/persistent malignancy requiring rapid immune suppression withdrawal.
* Active uncontrolled infection according to the attending physician
* Severe organ dysfunction unrelated to underlying GvHD, including:

Cholestatic disorders or unresolved veno-occlusive disease of the liver (defined as persistent bilirubin abnormalities not attributable to GvHD and ongoing organ dysfunction).

Clinically significant or uncontrolled cardiac disease including unstable angina, acute myocardial infarction within 6 months before Day 1 of study drug administration, New York Heart Association Class III or IV congestive heart failure, circulatory collapse requiring vasopressor or inotropic support, or arrhythmia that requires therapy.

Clinically significant respiratory disease that requires mechanical ventilation support or 50% oxygen.

* Current or past veno-occlusive disease or other uncontrolled complication unless otherwise agreed in writing by the sponsor.
* Absolute neutrophil count <500/µL for 3 consecutive days. Use of growth factor supplementation is allowed.
* Absolute platelet count < 10 000/µL. Use of platelet infusion is allowed.
* Patient with negative IgG EBV serology.
* Current or past evidence of toxic megacolon, bowel obstruction or gastrointestinal perforation.
* Any condition that would, in the investigator's judgment, interfere with full participation in the study, including administration of study drug and attending required study visits; pose a significant risk to the subject; or interfere with interpretation of study data.
* Known allergy or intolerance to trehalose or maltodextrin.
* Vulnerable patients such as: minors, persons deprived of liberty, persons in Intensive Care Unit unable to provide informed consent prior to the intervention.
* Females of childbearing potential should have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication. Females of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile or abstain from procreative sexual activity for the course of the study. Females of childbearing potential are those who have not been surgically sterilized or have not been free from menses for >1 year. Males should agree to abstain from procreative sexual activity starting with the first dose of study therapy through the end of the study.
* Other ongoing interventional protocol that might interfere with the current study's primary endpoint.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2022-03-25 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
ORR of gastro intestinal-aGvHD | Day 28
  Overall Response Rate (Complete Response + Very Good Partial Response + Partial Response)

SECONDARY OUTCOMES:
Safety and tolerability | Day 28
  Incidence of AEs, treatment-emergent AEs (TEAEs), Serious Adverse Events (SAEs), deaths, and laboratory abnormalities related to MaaT013, using the National Cancer Institute-Common Terminology Criteria for AEs (NCI-CTCAE) v5.0., and results from physical examination from D1 to Day 28.
Safety and tolerability | Month 3
  Incidence of AEs, treatment-emergent AEs (TEAEs), Serious Adverse Events (SAEs), deaths, and laboratory abnormalities related to MaaT013, using the National Cancer Institute-Common Terminology Criteria for AEs (NCI-CTCAE) v5.0.
Safety and tolerability | Month 12
  incidence of SAE and key events
aGvHD ORR | Day 28, Day 56 and Month 3
  aGvHD overall response rate (CR, VGPR and PR) for all organs
GI aGvHD ORR | Day 56 and Month 3
  GI aGvHD overall response rate (CR, VGPR and PR)
Best response rates | until Month 3
  CR, VGPR and PR for GI and overall aGvHD
Survival rates | Month and Month12
  Progression-free survival, relapse-free survival, overall survival, steroid-free survival, immunosuppression-free survival
Duration of response | Month 12
  Duration of response after D28
chronic GvHD incidence and severity | Month 12
  Percentage of chronic GvHD incidence and severity

OTHER OUTCOMES:
Exploratory endpoint | Day 28
  Evaluation of MaaT013 impact on blood GvHD immune markers

CONTACTS AND LOCATIONS:
Overall Officials: Florent Malard, MD, PhD, Principal Investigator — APHP
Locations (50):
- Austria (2):
  - Medizinische Universität Innsbruck, Innsbruck
  - Ordensklinikum Linz Elisabethinen, Linz
- Belgium (5):
  - Algemeen Ziekenhuis Sint-Jan Brugge-Oostende - Campus Sint-Jan, Bruges
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Brussel, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - Centre Hospitalier Universitaire de Liège, Liège
- France (16):
  - Centre Hospitalier Universitaire Amiens-Picardie - Site Sud, Amiens
  - Centre Hosptitalier Universitaire d'Angers, Angers
  - CHU de Caen, Caen
  - Centre Hospitalier Universitaire Grenoble Alpes, Grenoble
  - CHRU Lille - Hopital Claude Huriez, Lille
  - Institut Paoli Calmettes, Marseille
  - Hôpital Lapeyronie, Montpellier
  - Hôpital l'Archet, Nice
  - APHP St Antoine, Paris
  - Hôpital Haut-Lévêque, Pessac
  - Centre Hospitalier Lyon-Sud, Pierre-Bénite
  - Centre Hospitalier Universitaire de Poitiers, Poitiers
  - Hôpital Pontchaillou, Rennes
  - Institut de Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez
  - Institut Universitaire du Cancer de Toulouse Oncopole, Toulouse
  - Hôpitaux de Brabois, Vandœuvre-lès-Nancy
- Germany (5):
  - Helios Klinikum Berlin-Buch, Berlin
  - Universitätsmedizin Mannheim, Mannheim
  - Universitätsklinikum Regensburg, Regensburg
  - Universitätsklinik Ulm - Oberen Eselsberg, Ulm
  - Universitatsklinikum Wurzburg, Würzburg
- Italy (9):
  - Azienda Ospedaliera Regionale San Carlo, Ancona
  - Azienda Ospedaliero-Universitaria di Bologna Policlinico Sant Orsola-Malpighi, Bologna
  - Istituto di Ricovero e Cura a Carattere Scientifico - Ospedale Policlinico San Martino, Genova
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - IRCCS Ospedale San Raffaele, Milan
  - Grande Ospedale Metropolitano Bianchi Melacrino Morelli, Reggio Calabria
  - Fondazione Policlinico Universitario Agostino Gemelli, Roma
  - Azienda Ospedaliero-Universitaria Citta della Salute e della Scienza di Torino, Torino
  - Presidio Ospedaliero Universitario Santa Maria della Misericordia, Udine
- Spain (13):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Institut Català d'Oncologia - Hospital Duran i Reynals (ICO L'Hospitalet), Barcelona
  - Hospital Clínico Universitario Virgen de la Arrixaca, El Palmar
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital General Universitario Morales Meseguer, Murcia
  - Clinica Universidad de Navarra - Pamplona, Pamplona
  - Complejo Asistencial Universitario de Salamanca - Hospital Clínico, Salamanca
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Instituto de Biomedicina de Sevilla, Seville
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitari i Politècnic La Fe, Valencia

IPD SHARING:
Plan to Share IPD: Undecided